CLINICAL TRIAL: NCT00837343
Title: An Open Label, Multicenter, Single Arm, 4-Week Study to Evaluate the Efficacy and Safety of Flexible Dose of Quetiapine Fumarate (Seroquel) Switching From Other Drugs in the Treatment of Acute Manic Patients With Bipolar Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of Flexible Dose of Quetiapine Fumarate (Seroquel) Switching From Other Drugs in the Treatment of Acute Manic Patients With Bipolar Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Mental Hospital (Other)
Collaborators: First Affiliated Hospital of Jinan University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Guangzhou mental Hospital Attached to Guangzhou Civil Affairs Bureau (Unknown)
Responsible Party: Jie Li, Guangzhou Mental hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00070
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quetiapine Fumarate arm (Experimental): Quetiapine Fumarate arm
  Interventions: Drug: quetiapine fumarate tablet (Seroquel)

INTERVENTIONS:
Drug: quetiapine fumarate tablet (Seroquel) — Investigational product: quetiapine fumarate tablet (Seroquel) , 25 mg, 200 mg, 300mg, manufactured by AstraZeneca.The total daily doses of quetiapine fumarate will be increased to 600mg/d on the 6th since enrolment day. At day 7 or later, the dose can be adjusted in the range of 400- 800mg/day.

SUMMARY:
Bipolar disorder (BD) is also named as a bipolar affective disorder, belonging to a kind of severe mental disorder involving both mania or hypomania and depression episode, with lifetime prevalence between 1.2 - 1.6%. The hygienic burden of bipolar disorder is high, and its disease burden lies in top 10 position among the population of 15 - 44 years of old patients and concomitant with relative high suicide rate (10 - 15%) and mutilation rate, as reported by the World Health Organization (WHO) 2001 Annual Report. Drug treatment is one of the main treatment methods for this kind of disease, and the dose selected will interfere the efficacy and prognosis of the patient.

Quetiapine fumarate (Seroquel) is a dibenzothiazepine derivative, which is widely used in the world. It has the indications in schizophrenia, bipolar mania and depression approved by FDA. Quetiapine fumarate has been used in China for almost 10 years, which is in the treatment of schizophrenia. The indication of bipolar mania has been approved by SFDA recently. Exploration of the relationship between the dose and efficacy has been a hot spot in the clinical practice as the drug has a broad action spectrum and wide dose range (200mg/d-800mg/d).

Brain-derived neurotrophic factor (BDNF) plays an important role in the pathophysiology of bipolar disorder. Some clinical studies indicate the blood BDNF level decreased during the depression phase in the bipolar disorder, and the blood BDNF level is negative proportional to the severity of the depression; and the same phenomenon was found, i.e. the blood BDNF level decreased during the manic phase in the bipolar disorder, and the blood BDNF level is negative proportional to the severity of the mania. Quetiapine fumarate was found to reduce the decreasing of the expression of BDNF in the rat hippocampus and brain mantle in some animal experiments, indicating quetiapine fumarate has the possibility on potential interfering BDNF in the treatment. However, few study on comparison of the blood BDNF level between pre and post treatment in the bipolar disorder was conducted.

DETAILED DESCRIPTION:
This is a multicenter, open label, 4-week study. Study subjects are defined in Chinese Han nationality patients with acute mania of bipolar disorder (inpatients or outpatients). The screening phase is up to 7 days. The eligible patients in the screening phase can be enrolled into the treatment phase, the target dose is 400-800mg/day, and treatment period will last for 4 weeks. The objective is to evaluate the efficacy of quetiapine fumarate switching from other drugs used as monotherapy in the treatment of acute mania with bipolar disorder, and the relationship between the serum BDNF and quetiapine fumarate.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent was submitted by subjects or their legal guardian
2. Bipolar disorder (296.0x, 296.4x) is diagnosed by the Structured Clinical Interview for DSM-IV Axis I Disorders - Patient Edition (SCID), based on the 4th edition of US Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)
3. Aged between 18 and 65, male and female, Han nationality
4. In the acute phase of mania episode and YMRS total score is at least 22 at baseline.
5. The following drugs (lithium carbonate, sodium valproate, risperidone or olanzapine) were received as previous maintain treatment( monotherapy or combination therapy) in adequate dose according to label within three months before this mania episode.
6. Child-bearing potential female patients should conduct urine pregnancy test (HCG) at the enrolment, and the result should be negative; and also willing to take contraception measures during the study period
7. Be able to understand and comply with the requirements of the study

Exclusion Criteria:

1. Women in pregnancy or lactation
2. The duration of this mania episode is at most 2 weeks at enrollment.
3. DSM-IV Axis I Disorders except bipolar disorder (296.0x, 296.4x)
4. Patients with symptoms of obvious suicide (MADRS No. 10 score ≥4), self-injured or harmful to others, as judged by the investigators
5. Known intolerance or lack of response to quetiapine fumarate, as judged by the investigators
6. Patients with non-compliance by his history as judged by the investigators
7. Use of any potent cytochrome P450 3A4 inhibitors in the 14 days preceding randomization, including but not limited as ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine, and saquinavir
8. Use of potent cytochrome P450 inducers in the 14 days preceding randomization, including but not limited as phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
9. long-acting antipsychotic drug was injected within 1 injection interval (prolonged acting injection) before randomization
10. Use of clozapine in the 28 days preceding randomization
11. Substance or alcohol dependence according to the DSM-IV criteria at randomization (except complete recovered, and caffeine and nicotine dependence)
12. Dependence for the following drugs according to the DSM-IV standard at 4 weeks preceding randomization: opioids, amphetamine, barbiturates, cocaine, cannabis, or hallucinogens
13. Medical conditions that would affect absorption, distribution, metabolism or excretion of study treatment.
14. Clinical evidence for the relevant diseases (e.g. renal or hepatic dysfunction, severe coronary heart disease, cerebrovascular disease, hepatitis and acquired immunodeficiency syndrome (AIDS))
15. Unstable conditions (e.g. hypertension, congestive heart failure, unstable angina pectoris) or in the opinion of the investigator would be negatively affected by study medication or that would affect study medication, or has a medical history of chronic body disease.
16. Medical history with seizure disorder, except for febrile convulsion
17. Persons involved in the study design and conducting (suitable for the working staff in AstraZeneca and study site)
18. Participation in another clinical study within 4 weeks (or longer time according to the local requirement) of randomisation
19. Patients with diabetes mellitus (DM)
20. An absolute neutrophil count (ANC) of < 1.5 x 109/L
21. Thyroid-stimulating hormone level is more than 10% above the upper limit of the normal range, regardless of treatment for hypothyroidism or hyperthyroidism.
22. Abnormal ECG with clinical significance at enrollment indicating abnormal function in the heart, as judged by the investigator
23. Previous enrolment in the present study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy variable for this study is the YMRS total score change from baseline to Day 28 (LOCF). | 28 days

SECONDARY OUTCOMES:
To evaluate the effectiveness of quetiapine fumarate | 28 days
To evaluate the relationship between the serum brain-derived neurotrophic factor and quetiapine fumarate | 28 days
To evaluate the safety and tolerability of quetiapine fumarate | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, Professor, Principal Investigator — Guangzhou Mental Hospital
Locations (1):
- Guangzhou Mental Hospital, Guangzhou, China/Guangdong Province, China